CLINICAL TRIAL: NCT05037604
Title: Factors Associated With Dermatoporosis
Acronym: FAWD
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Director, Universidad Autonoma de San Luis Potosí
Other Study IDs: FactorsDermatoporosis
Record Dates: First submitted 2021-08-23; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Senile Purpura
Keywords: dermatoporosis; senile; purpura
MeSH Terms: conditions — Purpura | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients diagnosed with dermatoporosis. A clinical history, physical examination, and application of a previously validated diagnostic self-questionnaire were performed.
  Interventions: Other: Questionnaire about associated factors; Diagnostic Test: Self questionnaire diagnostic tool; Other: Physical Examination
- Control: Patients not diagnosed with dermatoporosis. A clinical history, physical examination, and application of a previously validated diagnostic self-questionnaire were performed.
  Interventions: Other: Questionnaire about associated factors; Diagnostic Test: Self questionnaire diagnostic tool; Other: Physical Examination

INTERVENTIONS:
Other: Questionnaire about associated factors — Questionnaire about age, prolonged sun exposure, intake of anticoagulants / antiplatelets, intake of oral steroids, chronic kidney disease. Maternal age> 40 years in their last child , time of lactation per pregnancy and cumulative time of lactation. Age of the first pregnancy and age of menopause onset.
Diagnostic Test: Self questionnaire diagnostic tool — Self questionnaire of physical characteristics
Other: Physical Examination — Physical Examination made by a dermatologist

SUMMARY:
Dermatoporosis is a chronic syndrome of skin insufficiency or fragility. It is characterized by cutaneous atrophy, senile purpura and stellate pseudoscars. Dermatoporosis prevalence is 37% in ≥65 years.

The objective was to determine factors associated with this diagnosis in >60 years old patients of the outpatient clinic in the Hospital Central "Dr. Ignacio Morones Prieto " San Luis Potosí, México.

An observational, cross-sectional, descriptive, and analytical study was performed. Patients >60 years old were selected. A clinical history, clinical examination, and application of a validated diagnostic self-questionnaire were performed.

DETAILED DESCRIPTION:
Dermatoporosis is a chronic syndrome of skin insufficiency or fragility. It is characterized by cutaneous atrophy, senile purpura and stellate pseudoscars. Dermatoporosis prevalence is 37% in ≥65 years.The objective was to determine factors associated with this diagnosis in >60 years old patients of the outpatient clinic in the Hospital Central "Dr. Ignacio Morones Prieto " San Luis Potosí, México.

An observational, cross-sectional, descriptive and analytical study was performed. Through consecutive non-probabilistic sampling, patients > 60 years old were selected, who underwent a clinical history, clinical examination, and the application of a validated diagnostic self-questionnaire. To determine the association of the factors, a multivariate logistic regression analysis, it will be used the PRIMERv6 software with the PERMANOVA package. A p <0.05 was considered significant. The normality of the distribution of the continuous variables was evaluated with the Shapiro Wilk test. The Student's t test was performed on variables that met the homogeneity of variance requirements. In the variables that did not meet this criterion, a non-parametric analysis was performed with the Mann U Whitney test. For the analysis of categorical variables, Fisher's exact test or chi-square test was used. Continuous variables were reported by mean (median) [Q1, Q3] (min - max) and by standard deviations as their distribution corresponds. Nominal categorical variables were expressed as frequencies

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years

Exclusion Criteria:

* Patients in whom physical examination cannot be performed due to the use of orthopedic devices such as splints, bandages, etc.
* Patients with whom interviewer-patient verbal communication is difficult due to some hearing or neurological deficit.
* Patients with neurological, psychiatric disorders who are unable to provide reliable information. (disorganized, incoherent speech, cognitive deficit)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years of age who attended the outpatient clinic of the Hospital Central "Dr. Ignacio Morones Prieto "
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Factors associated with Dermatoporosis | At time of enrollment
  Presence of factors related to age, sex, personal history of diseases, chronic oral treatments, gyneco-obstetrics background, chronic photoexposure
Diagnostic by self assesment tool | At time of enrollment
  Diagnostic of dermatoporosis made by self assesment tool
Physical examination | At time of enrollment
  Presence of pseudoscars (stellate scars) in the physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Castanedo-Cazares, PhD, Principal Investigator — Universidad Autonoma de San Luis Potosí
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database of 315 patients diagnosed and not diagnosed with dermatoporosis will be shared for 3 years. It includes associated factors, physical examination and results of self assesment tool.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: The database will be shared with researchers who require it by means of a letter sent to the principle investigator justifying its use for research and attaching a letter that describes the privacy policy to safeguard the information contained in the database.

REFERENCES:
- [Result] Kaya G, Kaya A, Sorg O, Saurat JH. Dermatoporosis: a further step to recognition. J Eur Acad Dermatol Venereol. 2018 Feb;32(2):189-191. doi: 10.1111/jdv.14777. No abstract available. PMID 29465833
- [Result] Han A, Chien AL, Kang S. Photoaging. Dermatol Clin. 2014 Jul;32(3):291-9, vii. doi: 10.1016/j.det.2014.03.015. PMID 24891052
- [Result] Kaya G, Saurat JH. Dermatoporosis: a chronic cutaneous insufficiency/fragility syndrome. Clinicopathological features, mechanisms, prevention and potential treatments. Dermatology. 2007;215(4):284-94. doi: 10.1159/000107621. PMID 17911985
- [Result] Kluger N, Impivaara S. Prevalence of and risk factors for dermatoporosis: a prospective observational study of dermatology outpatients in a Finnish tertiary care hospital. J Eur Acad Dermatol Venereol. 2019 Feb;33(2):447-450. doi: 10.1111/jdv.15240. Epub 2018 Oct 1. PMID 30198583
- [Result] Vanzi V, Toma E. Recognising and managing age-related dermatoporosis and skin tears. Nurs Older People. 2018 Mar 23;30(3):26-31. doi: 10.7748/nop.2018.e1022. PMID 29569862
- [Result] Kattoor AJ, Pothineni NVK, Palagiri D, Mehta JL. Oxidative Stress in Atherosclerosis. Curr Atheroscler Rep. 2017 Sep 18;19(11):42. doi: 10.1007/s11883-017-0678-6. PMID 28921056
- [Result] Rapa SF, Di Iorio BR, Campiglia P, Heidland A, Marzocco S. Inflammation and Oxidative Stress in Chronic Kidney Disease-Potential Therapeutic Role of Minerals, Vitamins and Plant-Derived Metabolites. Int J Mol Sci. 2019 Dec 30;21(1):263. doi: 10.3390/ijms21010263. PMID 31906008
- [Result] Gilchrest BA, Blog FB, Szabo G. Effects of aging and chronic sun exposure on melanocytes in human skin. J Invest Dermatol. 1979 Aug;73(2):141-3. doi: 10.1111/1523-1747.ep12581580. PMID 88488
- [Result] Dekel N, Gnainsky Y, Granot I, Mor G. Inflammation and implantation. Am J Reprod Immunol. 2010 Jan;63(1):17-21. doi: 10.1111/j.1600-0897.2009.00792.x. PMID 20059465
- [Result] Mor G. Inflammation and pregnancy: the role of toll-like receptors in trophoblast-immune interaction. Ann N Y Acad Sci. 2008 Apr;1127:121-8. doi: 10.1196/annals.1434.006. PMID 18443339
- [Result] Michaud M, Balardy L, Moulis G, Gaudin C, Peyrot C, Vellas B, Cesari M, Nourhashemi F. Proinflammatory cytokines, aging, and age-related diseases. J Am Med Dir Assoc. 2013 Dec;14(12):877-82. doi: 10.1016/j.jamda.2013.05.009. Epub 2013 Jun 20. PMID 23792036
- [Result] Straub RH, Schradin C. Chronic inflammatory systemic diseases: An evolutionary trade-off between acutely beneficial but chronically harmful programs. Evol Med Public Health. 2016 Jan 27;2016(1):37-51. doi: 10.1093/emph/eow001. PMID 26817483
- [Result] Ayala A, Munoz MF, Arguelles S. Lipid peroxidation: production, metabolism, and signaling mechanisms of malondialdehyde and 4-hydroxy-2-nonenal. Oxid Med Cell Longev. 2014;2014:360438. doi: 10.1155/2014/360438. Epub 2014 May 8. PMID 24999379
- [Result] Birben E, Sahiner UM, Sackesen C, Erzurum S, Kalayci O. Oxidative stress and antioxidant defense. World Allergy Organ J. 2012 Jan;5(1):9-19. doi: 10.1097/WOX.0b013e3182439613. Epub 2012 Jan 13. PMID 23268465
- [Result] Epel ES, Lithgow GJ. Stress biology and aging mechanisms: toward understanding the deep connection between adaptation to stress and longevity. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1(Suppl 1):S10-6. doi: 10.1093/gerona/glu055. PMID 24833580
- [Result] Butte NF, Hopkinson JM, Mehta N, Moon JK, Smith EO. Adjustments in energy expenditure and substrate utilization during late pregnancy and lactation. Am J Clin Nutr. 1999 Feb;69(2):299-307. doi: 10.1093/ajcn/69.2.299. PMID 9989696
- [Result] Mengeaud V, Dautezac-Vieu C, Josse G, Vellas B, Schmitt AM. Prevalence of dermatoporosis in elderly French hospital in-patients: a cross-sectional study. Br J Dermatol. 2012 Feb;166(2):442-3. doi: 10.1111/j.1365-2133.2011.10534.x. Epub 2011 Dec 5. No abstract available. PMID 21787367
- See also: INEGI. Población. Censos y conteos Población y Vivienda — https://www.inegi.org.mx/contenidos/productos/prod_serv/contenidos/espanol/bvinegi/productos/nueva_estruc/AEGEUM_2018/702825107000.pdf
- See also: ADULTOS MAYORES Análisis Integral de su Situación Jurídica en México — http://www.diputados.gob.mx/sedia/sia/spi/SAPI-ISS-11-17.pdf
- See also: Estimación del tiempo de exposición solar para quemadura en población mexicana. — https://www.medigraphic.com/cgi-bin/new/resumen.cgi?IDARTICULO=35548
- See also: INEGI. Encuesta Intercensal 2015 — https://www.inegi.org.mx/contenidos/productos/prod_serv/contenidos/espanol/bvinegi/productos/nueva_estruc/AEGEUM_2018/702825107000.pdf